CLINICAL TRIAL: NCT00872612
Title: Endosonography (EUS and EBUS) vs Conventional Bronchoscopy for the Diagnosis of Sarcoidosis: a Randomized Trial
Brief Title: Trial for the Diagnosis of Sarcoidosis
Acronym: GRANULOMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, M.B. von Bartheld, MB von Bartheld, MSc. PhD Student, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LUMC-GRANULOMA
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; Diagnosis; Non-caseating granulomas; BAL; EUS-FNA; EBUS-TBNA; TBLB
MeSH Terms: conditions — Sarcoidosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Endosonography arm
  Interventions: Procedure: EUS-FNA/EBUS-TBNA + BAL
- B (Active Comparator): Conventional bronchoscopy arm
  Interventions: Procedure: EBB + TBLB + BAL

INTERVENTIONS:
Procedure: EUS-FNA/EBUS-TBNA + BAL — EUS-FNA = Endoscopic Ultrasound guided fine needle aspiration of mediastinal lymph nodes.
  EBUS-TBNA = Endobronchial Ultrasound guided transbronchial needle aspiration of mediastinal and hilar lymph nodes.
  BAL = bronchoalveolar lavage
  Arms: A
Procedure: EBB + TBLB + BAL — EBB = Endobronchial biopsy TBLB = Transbronchial biopsy BAL = Bronchoalveolar lavage
  Arms: B

SUMMARY:
This randomized study investigates two different diagnostic strategies for patients with suspected pulmonary sarcoidosis stage I/II.

The objective is to assess the role of endosonography (EBUS/ EUS - FNA) in demonstrating non-caseating granulomas in comparison with conventional bronchoscopy (TBLB + EBB).

Also the researchers investigate the additional value of BAL, in relation to endosonography and conventional bronchoscopy (TBLB + EBB), in diagnosing sarcoidosis.

Thirdly the researchers aim to assess the rate of complications in both the endosonography and conventional bronchoscopic workup.

DETAILED DESCRIPTION:
Sarcoidosis is the most prevalent interstitial lung disease in Western-Europe and the US. The disease is most prevalent in young adults. To set the final diagnosis of sarcoidosis, the following parameters need to be present:

1. A clinical and radiological suspicion of sarcoidosis stage I/II.
2. A tissue diagnosis of disease-specific non-caseating granulomas.
3. Exclusion of possible alternative diagnoses as lung cancer or tuberculosis.

Nowadays, a bronchoscopy with lung biopsies is advised to set a tissue diagnosis of sarcoidosis. However, these biopsies are only diagnostic in 70% of the procedures and they are associated with a 3% risk of coughing up blood and a 4% risk of a lung collapse.

Since recently, a new diagnostic procedure has come available. This procedure, endo-sonography, makes it possible to biopsy lymph nodes in the chest under direct visualization and has a diagnostic accuracy of 85%. The associated risk of complications appears to be small (<1%)

We consider the current standard for the diagnostics of sarcoidosis to be outdated, considering the clinical availability of endo-sonography. We expect that endo-sonography is more frequent diagnostic for a tissue diagnosis of sarcoidosis.

Also we hypothesize that this technique is safer and more preferred by patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected pulmonary sarcoidosis stage I/ II
* Age > 18 years
* Both males and females
* Written informed consent is obtained.

Exclusion Criteria:

* Patients with obvious other organ involvement of sarcoidosis where a simple diagnostic biopsy to assess granulomas can be performed.
* Löfgren's syndrome
* Inability to undergo fiberbronchoscopy, EBUS or EUS (e.g. respiratory insufficiency, esophageal stenosis
* Contraindications for a lung or nodal biopsy (e.g. coagulopathy, thrombocytopenia)
* Pregnancy
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The role of endosonography (EBUS/ EUS - FNA) in demonstrating non-caseating granulomas in comparison with conventional bronchoscopy (TBLB + EBB) | within a week

SECONDARY OUTCOMES:
Assessment of complications of both the endosonography and conventional bronchoscopic workup | within 30 days
The additional value of BAL, in relation to endosonography and conventional bronchoscopy (TBLB + EBB), in diagnosing sarcoidosis | 2 weeks
Assessment of patient preference for both the endosonographic and conventional bronchoscopic work-up. | within a week

CONTACTS AND LOCATIONS:
Overall Officials: M B von Bartheld, MSc, Study Director — Pulmonary Department, Leiden University Medical Center; J T Annema, MD PhD, Principal Investigator — Pulmonary Department, Leiden University Medical Center; K F Rabe, MD PhD, Principal Investigator — Pulmonary Department, Leiden University Medical Center
Locations (15):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Gentofte Hospital Copenhagen, Hellerup, Copenhagen, Denmark
- Germany (2):
  - Thoraxklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Hospital Grosshansdorf, Großhansdorf, Schleswig-Holstein
- Netherlands (7):
  - Rijnstaete Ziekenhuis, Arnhem, Gelderland
  - Radboud Universitair Medisch Centrum, Nijmegen, Gelderland
  - St. Catharina Ziekenhuis, Eindhoven, North Brabant
  - Pulmonary Department, Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - St. Franciscus Ziekenhuis, Rotterdam, South Holland
  - Medisch Centrum Haaglanden, The Hague, South Holland
- Poland (2):
  - University hospital Krakow, J.P. II, Krakow
  - Sokołowski Pulmonary Hospital, Zakopane
- United Kingdom (2):
  - Royal Brompton Hospital, London, London
  - Chelsea and Westminster hospital, London

REFERENCES:
- [Background] Costabel U, Hunninghake GW. ATS/ERS/WASOG statement on sarcoidosis. Sarcoidosis Statement Committee. American Thoracic Society. European Respiratory Society. World Association for Sarcoidosis and Other Granulomatous Disorders. Eur Respir J. 1999 Oct;14(4):735-7. doi: 10.1034/j.1399-3003.1999.14d02.x. No abstract available. PMID 10573213
- [Background] Iannuzzi MC, Rybicki BA, Teirstein AS. Sarcoidosis. N Engl J Med. 2007 Nov 22;357(21):2153-65. doi: 10.1056/NEJMra071714. No abstract available. PMID 18032765
- [Background] Winterbauer RH, Lammert J, Selland M, Wu R, Corley D, Springmeyer SC. Bronchoalveolar lavage cell populations in the diagnosis of sarcoidosis. Chest. 1993 Aug;104(2):352-61. doi: 10.1378/chest.104.2.352. PMID 8339618
- [Background] Kantrow SP, Meyer KC, Kidd P, Raghu G. The CD4/CD8 ratio in BAL fluid is highly variable in sarcoidosis. Eur Respir J. 1997 Dec;10(12):2716-21. doi: 10.1183/09031936.97.10122716. PMID 9493649
- [Background] Annema JT, Veselic M, Rabe KF. Endoscopic ultrasound-guided fine-needle aspiration for the diagnosis of sarcoidosis. Eur Respir J. 2005 Mar;25(3):405-9. doi: 10.1183/09031936.05.00098404. PMID 15738281
- [Background] Garwood S, Judson MA, Silvestri G, Hoda R, Fraig M, Doelken P. Endobronchial ultrasound for the diagnosis of pulmonary sarcoidosis. Chest. 2007 Oct;132(4):1298-304. doi: 10.1378/chest.07-0998. Epub 2007 Sep 21. PMID 17890467
- [Derived] von Bartheld MB, Dekkers OM, Szlubowski A, Eberhardt R, Herth FJ, in 't Veen JC, de Jong YP, van der Heijden EH, Tournoy KG, Claussen M, van den Blink B, Shah PL, Zoumot Z, Clementsen P, Porsbjerg C, Mauad T, Bernardi FD, van Zwet EW, Rabe KF, Annema JT. Endosonography vs conventional bronchoscopy for the diagnosis of sarcoidosis: the GRANULOMA randomized clinical trial. JAMA. 2013 Jun 19;309(23):2457-64. doi: 10.1001/jama.2013.5823. PMID 23780458